CLINICAL TRIAL: NCT02663856
Title: My Smart Age With HIV (MySAwH): Smartphone Self-assessment of Frailty and Information - Communication Technology to Promote Healthy Ageing in HIV.
Brief Title: My Smart Age With HIV: Smartphone Self-assessment of Frailty
Acronym: MySAwH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Giovanni Guaraldi, MD, University of Modena and Reggio Emilia
Other Study IDs: MySAwH
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: HIV Infection; Aging
MeSH Terms: conditions — HIV Infections | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational — Self assessment of ageing transition using a frailty index through MySAwH app

SUMMARY:
Understanding the complexity of aging and frailty in chronic HIV infection motivated Italian team members to begin to build a frailty index (FI) including 37 health variables at the Modena HIV Metabolic Clinic (MHMC). The validation of FI in HIV patients have been recently published, and more data comparing FI in HIV infected vs un-infected people, have been presented at international meeting and are at present submitted for publication.

The research consortium (MHMC, HCC and HHMP) of this study was motivated to begin preliminary work in consideration of the similar multidisciplinary approach in Ageing care and capacity to address health status in ageing HIV patients using shared definitions of co-morbidities, multi-morbidity and measures of Physical Function and Cognition impairment, disability and quality of life. The investigators wanted to overcome the major criticism intrinsic in the FI, that is the needs to collects many variables not easily available in most HIV centres. The the investigators approach is to make patient living with HIV (PLWH), be the source of health variables taking advantage of information and communication technologies available with smart phones and fitness tracking device, collecting physiological parameters and patient related outcomes.

DETAILED DESCRIPTION:
In this study the investigators plan to empower elderly HIV patients via health promotion, assessing reduction in health deficit and improvement in quality of life using My Smart Age (MySAwH) application.

MySAwH is an interactive mobile application designed to empower elderly HIV patients in health promotion through self assessment of ageing transition using a FI. FI is generated from health variables which include physical function data routinely collected by fitness tracking devices, Ecological momentary assessment data collected with smart phones and Physician health data collected during patient visits. The change in frailty index over time describes health transition. Although health generally worsens with age, the relationship between aging and health is dynamic and periodic improvement and stability in frailty index may be the result of the patients engagement in health promotion and improved life style.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection on ART
* HIV1-RNA<40 c/mL for at least 6 months
* Age stratification:

  * 50 pts (per centre) aged 50-64 years
  * 50 pts (per centre) aged ≥ 65 years
* Routine access to a smart phone and willingness to use the fitness tracking device
* Willingness to be trained to use an interactive mobile application

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In a prospective 24 months study, 300 consecutive HIV positive patients aged>50 years (100 per centre)will be enrolled to assess primary objective.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Measure change of frailty index | 18 months
  Assed by MySAwH application
Measure Multi-morbidity | 18 months
  Assed by physician, based on the presence of 2 or more co-morbidities (hypertension, diabetes, cardiovascular disease, etc)
Measure Physical Function | 18 months
  Assed using a Short Physical Performance Battery
Measure Cognition impairment | 18 months
  Assed using neurocognitive tests
Measure disability | 18 months
  Assed using disability questionnaire
Measure quality of life | 18 months
  Assed using quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Guaraldi, Prof, Principal Investigator — University of Modena and ReggioEmilia
Locations (1):
- Clinica Metabolica, Ambulatorio HIV, A.O.U. Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No